CLINICAL TRIAL: NCT05930236
Title: Ultrasound-guided Medial Lumbar Bundle Branch Block by Caudal-cranial Approach: Radiographic Comparison of a New Ultrasound-guided Method
Brief Title: Ultrasound-guided LMBB by Caudal-cranial Approach: Radiographic Comparison of a New Ultrasound-guided Method
Acronym: BLEPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Marie-Laure Nisolle, Nisolle Marie-Laure, MD, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2023/034
Record Dates: First submitted 2023-06-22; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Chronic Low-back Pain; Lumbar Facet Joint Syndrome
Keywords: Pain; fluoroscopy; Ultrasound; Injection Site Infiltration; Chronic; facet infiltration
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Iohexol

STUDY DESIGN:
Intervention Model Description: the medial branch block on three lumbar levels (L3-L4, L4-L5 and L5-S1) will be performed under ultrasound by "caudal-cranial" approach, followed by an X-ray check to verify the positioning of the needle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound guided infiltration verified by fluoroscopy (Experimental): The 22G needle is introduced along a caudal-cranial axis to infiltrate at each level a volume of 1mL of a mixture consisting of 3mL of Linisol 2% (60mg of lidocaine) and 1mL of Depomedrol (Methylprednisolone) 40mg with 1mL of Omnipaque (contrast product). At each level, contrast medium will be injected at the same time as the linisol-depomedrol mixture so that once the BBM under ultrasound is completed, an X-ray check is performed.
  Interventions: Diagnostic Test: Lumbar medial branch block; Drug: Lidocain; Drug: Methylprednisolone; Drug: Omnipaque

INTERVENTIONS:
Diagnostic Test: Lumbar medial branch block — The lumbar medial branch block on three lumbar levels (L3-L4, L4-L5 and L5-S1) will be performed by ultrasound-guidance in a longitudinal plane and the correct placement of the needle will be verified by radiography to show if the two modalities are equivalent.
  Other Names: LMBB
Drug: Lidocain — Linisol infiltration with depomedrol and omnipaque
  Other Names: linisol
Drug: Methylprednisolone — infiltration with linisol and omnipaque
  Other Names: solumedrol
Drug: Omnipaque — infiltration with linisol and methylprednisolone

SUMMARY:
The current standard technique is radiography requiring three uni- or bilateral punctures (transverse-axial plane). The ultrasound technique is also described mainly in this plan but a new "caudal-cranial" ultrasound-guided technique was described by Chang et al in 2018 in which the major axis is used to conduct the needle to the desired area. The investigators would like to confirm that this new technique in a single puncture is also possible under ultrasound.

DETAILED DESCRIPTION:
The convex probe is first positioned in the median longitudinal plane opposite the spinous processes of the lower lumbar vertebrae L4 and L5 with the coordinate system on the cranial side and the side opposite the mark on the sacrum side. The latter is visualized as a hyperechogenic continuous line. The probe is then moved away from the midline, the probe is slightly inclined in an oblique paramedian position looking towards the midline, and gradually slid towards laterality in order to reveal successively, the plane of the laminar interlines of the L3, L4 and L5 vertebrae, then the plane of the facelet spacing of these same vertebrae at the junction of the upper and lower articular processes, finally the plane of their transverse processes

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain compatible with facet lumbar syndrome with chronic pain of at least 3 months
* who have not responded to conservative treatment after at least 4 weeks
* patients without signs of dissociated pain, radiculitis, neurological diseases including stroke and Parkinson's disease, spinal instability or deformities such as scoliosis, ankylosing spondylitis, history of lumbar surgery, fracture or lumbar tumor

Exclusion Criteria:

* Pregnant or breastfeeding women
* Allergy to injected products (Depomedrol or Linisol)
* Psychiatric disorders hindering understanding of the protocol
* Local or systemic infection
* Coagulation disorder
* Obese with a BMI> 35 kg / m²

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Correct needle placement rate | 0 min
  Check the correct placement of the needle placed by caudal-cranial approach by X-ray to show if the placement is correct (at the same time)

SECONDARY OUTCOMES:
change in visual analog scale (VAS) pain score | 30 min
  from baseline to 30 min after infiltration. scale (0 = no pain; 10 = worst pain imaginable)
Incidence of Adverse event | 30 min
  (Hematoma, infection, intrathecal injection, spinal anesthesia)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No